CLINICAL TRIAL: NCT06009224
Title: The Effect of Enhanced Recovery After Surgery (ERAS) on Pancreaticoduodenectomy in Patients With Hepatobiliary-Pancreas (HBP) Disease
Brief Title: The Effect of ERAS on Pancreaticoduodenectomy (v2.0)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae Wook Hwang, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1204
Record Dates: First submitted 2022-11-16; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Periampullary Cancer; Borderline Malignancy Tumor
Keywords: Enhanced Recovery After Surgery; Pancreaticoduodenectomy; Periampullary cancer; Fast track surgery; Postoperative complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Two study groups (Control (conventional) group and study (intervention) group) were randomly allocated and assigned to one of two groups in parallel for the whole duration of this study.
Who Masked: Outcomes Assessor
Masking Description: The evaluation and judgment for morbidity (primary endpoint) / mortality (secondary endpoint) was made by Morbidity and Mortality Committee in our division. Committee members were blinded about knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): Conventional ERAS program
- Experimental (Experimental): complete ERAS program (Conventional ERAS program + Epidural analgesia + Fluid balance)
  Interventions: Other: ERAS perioperative management

INTERVENTIONS:
Other: ERAS perioperative management — * Epidural analgesia
  * Fluid balance
  * Other items are the same as conventional
  Other Names: Fast tract
  Arms: Experimental

SUMMARY:
Enhanced Recovery After Surgery (ERAS) is not a program that aims to reduce postoperative hospital stay, but the multimodal strategies that aim to attenuate the loss of, and improve the restoration of, functional capacity after surgery on evidence-based medicine. The benefits of ERAS are proven in many surgical procedures, such as upper gastrointestinal surgery and colorectal surgery.

Investigators performed Randomized Controlled Trials to evaluate the non-inferiority of modified ERAS protocol for pancreaticoduodenectomy (PD) by introducing standardized pre- and post-operative treatment based on ERAS treatment guidelines (ERAS on PD, Research Institute Clinical Progress, 2014-0961; ClinicalTrials.gov, NCT02372331). As a result of the study, the ERAS protocol proved to be non-inferior to the existing pre- and post-operative treatment in terms of surgical complications, mortality, hospital stay, total hospital cost, and most nutritional indicators.

However, the previous study did not include a few important intraoperative items such as epidural analgesia and fluid balance among the main items of the ERAS protocol. This trial aims to evaluate the clinical results by applying the complete ERAS protocol.

DETAILED DESCRIPTION:
This study was a single-institution, randomized controlled clinical trial to test the superiority of Enhanced Recovery After Surgery (ERAS) protocol for patients with pancreaticoduodenectomy (PD).

This study will be conducted on adult patients who are planning to undergo pancreaticoduodenectomy for the treatment of periampullary disease for 12 months after the start of the study.

Based on the results of the previous study which choose the functional recovery date as a primary outcome (control group; 9.0 ± 4.3 days, intervention group; 7.6 ± 4.3 days), a total of 334 patients (167 patients in each group) will be enrolled when calculated with power 0.8, α = 0.05, a two-tailed test, and a 10% withdrawal rate.

Investigators plan to randomize patients covered by the existing ERAS program to the control group and patients covered by the full ERAS protocol to the experimental group.

Investigators plan to observe the clinical outcomes up to 3 months after surgery.

The primary outcome is the functional recovery date, and secondary outcomes are the postoperative complication rate, postoperative mortality, and readmission rate.

All subjects who were randomized and received any study intervention were obliged to follow the study protocol and monitored for best compliance, per-protocol set or safety set was not defined differently.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old
* Performance: Eastern Cooperative Oncology Group (ECOG) 0-2
* Resectable or borderline resectable malignant tumor or borderline malignant tumor on the periampullary area
* No distant metastases
* Bone marrow function: White Blood Cell (WBC) at least 3,000/mm3 or Absolute Neutrophil Count (ANC) ≥ 1,500/mm3, Platelet count at least 125,000/mm3
* Liver function: aspartate aminotransferase (AST) / alanine aminotransferase (ALT) less than 3 times the upper limit of normal
* Renal function: Creatinine no greater than 1.5 times the upper limit of normal
* Patients who consented and signed informed consent

Exclusion Criteria:

* Patients with distant metastases or patients with recurrent periampullary carcinoma
* Patients with active or uncontrolled infection
* Patients with severe psychiatric/neurological disorders
* People who are addicted to alcohol or other drugs
* Patients included in other clinical studies that may affect this study
* Patients unable to follow the researcher's instructions
* Pregnancy
* Patients with uncontrolled heart disease
* Patients with moderate or more comorbidities that are judged to have an impact on quality of life or nutritional status (liver cirrhosis, chronic renal failure, heart failure, etc.)
* Patients who underwent major abdominal organ surgery other than scheduled pancreaticoduodenectomy.
* Patients who require combined resection of other major abdominal organs in addition to scheduled pancreaticoduodenectomy
* History of allergy to local anesthetics
* Local infection at the treatment site
* Patients with neurological or mental health conditions
* A history of spinal surgery or compression fractures at abdominal level
* Patients with coagulopathy (Platelet < 125,000/mm3 or International Normalized Ratio (INR) ≥ 1.5) or who continue to take anticoagulants or antithrombotic drugs without stopping
* Others who are not suitable for research in the judgment of the clinician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional recovery date on postopreative 7th day | The investigators evaluate the five items to the participant starting on the 7th day after surgery. A date that satisfies all five items is defined as functional recovery date.
  * Pain control is possible only with oral or patch-type analgesics without intravenous analgesic administration
  * Able to walk freely
  * Free eating is possible
  * There should be no evidence of infection related to surgery
  * No intravenous nutritional injection (total parenteral nutrition) being administered

SECONDARY OUTCOMES:
Postoperative complication | Three months after surgery
  All complications after surgery are included. Especially, delayed gastric emptying, postpancreatectomy hemorrhage, postoperative pancreatic fistula and chyle leak will be classified by the criteria of International Study Group on Pancreatic Surgery.
  The severity of all complication will be divided depends on Clavien Dindo classification (Grade from I to V, higher scores mean a better outcome).
Postoperative mortality | 90 days after surgery
  All in-hospital mortality and 90 days mortality
Re-admission rate | 3 months after surgery
  For any reason, all readmitted patients are included.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Wook Hwang, M.D., PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It can be determined in accordance with the Personal Information Protection Act of KOREA and institutional data sharing regulations.

REFERENCES:
- [Result] Hwang DW, Kim HJ, Lee JH, Song KB, Kim MH, Lee SK, Choi KT, Jun IG, Bang JY, Kim SC. Effect of Enhanced Recovery After Surgery program on pancreaticoduodenectomy: a randomized controlled trial. J Hepatobiliary Pancreat Sci. 2019 Aug;26(8):360-369. doi: 10.1002/jhbp.641. Epub 2019 Jul 2. PMID 31152686
- [Result] Melloul E, Lassen K, Roulin D, Grass F, Perinel J, Adham M, Wellge EB, Kunzler F, Besselink MG, Asbun H, Scott MJ, Dejong CHC, Vrochides D, Aloia T, Izbicki JR, Demartines N. Guidelines for Perioperative Care for Pancreatoduodenectomy: Enhanced Recovery After Surgery (ERAS) Recommendations 2019. World J Surg. 2020 Jul;44(7):2056-2084. doi: 10.1007/s00268-020-05462-w. PMID 32161987
- [Result] Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, Gan TJ, Kennedy RH, Ljungqvist O, Lobo DN, Miller T, Radtke FF, Ruiz Garces T, Schricker T, Scott MJ, Thacker JK, Ytrebo LM, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice. Acta Anaesthesiol Scand. 2016 Mar;60(3):289-334. doi: 10.1111/aas.12651. Epub 2015 Oct 30. PMID 26514824
- [Result] Kuemmerli C, Tschuor C, Kasai M, Alseidi AA, Balzano G, Bouwense S, Braga M, Coolsen M, Daniel SK, Dervenis C, Falconi M, Hwang DW, Kagedan DJ, Kim SC, Lavu H, Liang T, Nussbaum D, Partelli S, Passeri MJ, Pecorelli N, Pillai SA, Pillarisetty VG, Pucci MJ, Su W, Sutcliffe RP, Tingstedt B, van der Kolk M, Vrochides D, Wei A, Williamsson C, Yeo CJ, Zani S, Zouros E, Abu Hilal M. Impact of enhanced recovery protocols after pancreatoduodenectomy: meta-analysis. Br J Surg. 2022 Feb 24;109(3):256-266. doi: 10.1093/bjs/znab436. PMID 35037019
- [Result] Lee JH, Kim DH, Koh WU. Real-time ultrasound guided thoracic epidural catheterization: a technical review. Anesth Pain Med (Seoul). 2021 Oct;16(4):322-328. doi: 10.17085/apm.21060. Epub 2021 Oct 29. PMID 34289297
- [Result] Kim HE, Kim YH, Song KB, Chung YS, Hwang S, Lee YJ, Park KM, Kim SC. Impact of critical pathway implementation on hospital stay and costs in patients undergoing pancreaticoduodenectomy. Korean J Hepatobiliary Pancreat Surg. 2014 Feb;18(1):14-20. doi: 10.14701/kjhbps.2014.18.1.14. Epub 2014 Feb 24. PMID 26155241